CLINICAL TRIAL: NCT05708911
Title: Impact of External Pharyngeal Exerciser on Pharyngeal Phase of Swallowing
Brief Title: External Pharyngeal Exerciser and Pharyngeal Phase of Swallowing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Reza Shaker, MD, Associate Provost for Clinical and Translational Research, Senior Associate Dean and Director of the Clinical and Translational Science Institute of SE WI, and the Joseph E. Geenen Professor and Chief of Gastroenterology and Hepatology, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00022959
Record Dates: First submitted 2023-01-13; First posted 2023-02-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Study of healthy subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Pharyngeal exerciser group (Experimental): Test that application of the pharyngeal exerciser increases the workload of muscles involved in pharyngeal phase of swallowing as evidenced manometrically by changes in
  Pharyngeal peak pressures Pharyngeal (velopharynx, oropharynx and hypopharynx) contractile duration Pharyngeal (velopharynx, oropharynx and hypopharynx) contractile integral Hypopharyngeal intrabolus pressure and duration UES nadir pressure UES relaxation time Baseline UES pressure
  Interventions: Device: Pharyngeal exerciser

INTERVENTIONS:
Device: Pharyngeal exerciser — Pharyngo-esophageal manometry during lateral fluoroscopy

SUMMARY:
This study of healthy young and elderly individuals is intended to assess the effects of pharyngeal exerciser on pharyngeal pressure phenomenon during swallowing. Our specific aim is to test if the pharyngeal exerciser increases the workload of muscles involved in pharyngeal phase of swallowing.

DETAILED DESCRIPTION:
1. All the study subjects are required to be without oral food or fluid intake for at least 3 hours prior to the study.
2. The participant's neck's physical dimensions and the device's physical dimensions will be measured and recorded. A physical examination including carotid artery auscultation will be performed.
3. After the application of local lidocaine, the high-resolution manometry (HRM) catheter will be inserted through the more patent nares and positioned such that it covers the entire pharynx from the nasopharynx to the proximal esophagus. In this position, manometry recording of the entire pharynx will be possible.
4. The pharyngeal exerciser will be placed around the neck overlying the larynx. The device will be in contact with the skin without any underlying pressure using the Velcro fastening in the back of the neck.
5. Patients will be sitting in an upright position and acclimatized for 10 minutes before proceeding.
6. Each subject will perform the following swallows:
7. Dry swallows x 5 times.

5 ml and 10 ml- of water swallows at room temperature x 5 times each.

5 ml and 10 ml- mashed potato swallowed at room temperature x 5 times each.

8. The sequence of the swallow types will be randomized. The swallow will be performed under device pressure of zero, 20, 30, 40 and 60 mm Hg in a randomized fashion. Each swallow type will be repeated 5 times with 30-second intervals in between.

9. The externally applied pressure will be measured by means of the pressure gauge included in the device

10. All the subjects will be given the option to participate in the concurrent videofluoroscopic examination along with pharyngeal manometry

11. The fluoroscopy machine will be turned "on" for 5 seconds only during the swallowing. The rest of the time fluoroscopy machine will be turned off.

12. These subjects undergoing concurrent fluoroscopy and manometry will perform the following swallows at zero, 20, and 40 mm Hg of device pressure:

Dry swallows x 3 times.

5 ml and 10 ml of water mixed barium swallow at room temperature x 3 times each.

5 ml- mashed potatoes mixed with barium at room temperature x 3 times.

The participant will also be instructed to resume their regular diet and activity.

All the tracings and video recordings will be analyzed by two individuals in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers must be at least 18 years of age or older.

Exclusion Criteria:

* Subjects with cervical spine disorders.
* Subjects with neurological disorders like dementia, cerebrovascular diseases other than Parkinson's Disease
* Subjects with carotid artery bruit or carotid vascular disorders.
* Subjects suffering from muscle diseases like muscular dystrophies, myopathies.
* Subjects with neuro-muscular junction disorders myasthenia gravis, Eaton-Lambert disorders.
* Subjects with any current esophageal symptoms like heartburn, dysphagia, chest pain or regurgitation.
* Subjects cannot have previous head or neck surgery or radiation.
* Subjects unable to tolerate nasal intubation.
* Subjects with significant bleeding disorders for whom nasal intubation has been deemed contraindicated.
* Subjects with a known upper airway or esophageal obstruction preventing the passage of the manometry probe.
* Subjects with autonomic dysfunction.
* Subjects having a history of allergy to lidocaine and barium.
* Subjects who are pregnant or lactating.
* Subjects who have advanced medical disorders (e.g.: chronic obstructive pulmonary disease (COPD), congestive heart failure, cirrhosis, cancer, chronic renal failure, etc.).
* Subjects who are medically unstable.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09-16 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
laryngeal excursion during swallowing | During mano-fluorography procedure
  maximum laryngeal excursion from resting position measured from fluoroscopic images during swallowing
hyoid excursion during swallowing | During mano-fluorography procedure
  maximum hyoid bone excursion from resting position measured from fluoroscopic images during swallowing
upper esophageal sphincter (UES) opening during swallowing | During mano-fluorography procedure
  maximum UES anterior-posterior diameter measured from fluoroscopic images during swallowing
pharyngeal peak peristaltic pressure | During mano-fluorography procedure
  maximum deglutitive pressure within the pharynx
pharyngeal (velopharynx, oropharynx and hypopharynx) contractile duration | During mano-fluorography procedure
  manometric duration of peristaltic pressure wave in velopharynx, oropharynx and hypopharynx
pharyngeal (velopharynx, oropharynx and hypopharynx) contractile integral | During mano-fluorography procedure
  space-time and length integral of pharyngeal pressures in the velopharynx, oropharynx and hypopharynx
hypopharyngeal intrabolus pressure | During mano-fluorography procedure
  maximum pressure within the hypopharynx as the swallowed bolus covers the pressure sites within the hypopharynx
hypopharyngeal intrabolus duration | During mano-fluorography procedure
  duration of maximum pressure within the hypopharynx as the swallowed bolus covers the pressure sites within the hypopharynx
UES nadir pressure | During mano-fluorography procedure
  minimum pressure within the upper esophageal sphincter (UES) during UES deglutitive relaxation
UES relaxation time | During mano-fluorography procedure
  duration pressure drops within the upper esophageal sphincter during UES deglutitive relaxation
baseline UES pressure | During mano-fluorography procedure
  average UES pressure when no swallow activity is present

CONTACTS AND LOCATIONS:
Overall Officials: Reza Shaker, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No